CLINICAL TRIAL: NCT03651128
Title: A Phase 3, Multicenter, Randomized, Open-label Study to Compare the Efficacy and Safety of bb2121 Versus Standard Regimens in Subjects With Relapsed and Refractory Multiple Myeloma (RRMM) (KarMMa-3)
Brief Title: Efficacy and Safety Study of bb2121 Versus Standard Regimens in Subjects With Relapsed and Refractory Multiple Myeloma (RRMM)
Acronym: KarMMa-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB2121-MM-003; U1111-1217-9988 (Registry Identifier: WHO); 2018-001023-38 (EudraCT Number)
Record Dates: First submitted 2018-08-16; First posted 2018-08-29 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; bb2121; Relapsed and Refractory Multiple Myeloma; High Risk Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — idecabtagene vicleucel; daratumumab; pomalidomide; Dexamethasone; Bortezomib; ixazomib; Lenalidomide; carfilzomib; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Administration of bb2121 (Experimental): bb2121 autologous CAR T cells will be infused at a dose ranging from 150 - 450 x 10^6 CAR+ T cells after receiving lymphodepleting chemotherapy
  Interventions: Biological: bb2121
- Arm B- standard regimens as per Investigator's discretion (Experimental): The participants will receive one of following regimens dependent on the subject's most recent anti-myeloma treatment regimen:
  * Daratumumab (DARA) in combination with pomalidomide (POM) and low-dose dexamethasone (dex) (DPd) OR
  * DARA in combination with bortezomib (BTZ) and low-dose dex (DVd) OR
  * Ixazomib (IXA) in combination with lenalidomide (LEN) and low-dose dex (IRd) OR
  * Carfilzomib (CFZ) in combination with low-dose dexamethasone (Kd) OR
  * Elotuzumab (ELO) in combination with POM and low-dose dexamethasone (EPd)
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib; Drug: Ixazomib; Drug: Lenalidomide; Drug: Carfilzomib; Drug: Elotuzumab

INTERVENTIONS:
Biological: bb2121 — bb2121
  Arms: Arm A - Administration of bb2121
Drug: Daratumumab — Daratumumab
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Pomalidomide — Pomalidomide
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Dexamethasone — Dexamethasone
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Bortezomib — Bortezomib
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Ixazomib — Ixazomib
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Lenalidomide — Lenalidomide
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Carfilzomib — Carfilzomib
  Arms: Arm B- standard regimens as per Investigator's discretion
Drug: Elotuzumab — Elotuzumab
  Arms: Arm B- standard regimens as per Investigator's discretion

SUMMARY:
This is a multicenter, randomized, open-label, Phase 3 study comparing the efficacy and safety of bb2121 versus standard regimens in subjects with relapsed and refractory multiple myeloma (RRMM).

The study is anticipated to randomize approximately 381 subjects with RRMM. Approximately 254 subjects will be randomized to Treatment Arm A and approximately 127 subjects will be randomized to Treatment Arm B.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements within this protocol and for a subject randomized to Treatment Arm A, subject agrees to continued follow-up for up to 15 years as mandated by the regulatory guidelines for gene therapy trials.
4. Subject has documented diagnosis of MM and measurable disease, defined as:

   * M-protein (serum protein electrophoresis [sPEP] or urine protein electrophoresis [uPEP]): sPEP ≥ 0.5 g/dL or uPEP ≥ 200 mg/24 hours and/or
   * Light chain MM without measurable disease in the serum or urine: Serum immunoglobulin free light chain ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa lambda free light chain ratio
5. Subject has received at least 2 but no greater than 4 prior MM regimens.
6. Subject has received prior treatment with DARA, a proteasome inhibitor- and an immunomodulatory compound-containing regimen for at least 2 consecutive cycles.
7. Subject must be refractory to the last treatment regimen. Refractory is defined as documented progressive disease during or within 60 days (measured from the last dose of any drug within the regimen) of completing treatment with the last anti-myeloma regimen before study entry.
8. Subject achieved a response (minimal response [MR] or better) to at least 1 prior treatment regimen.
9. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Recovery to Grade 1 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 2 peripheral neuropathy.
11. Adequate vascular access for leukapheresis
12. Females of childbearing potential (FCBP) must:

    a. Have negative pregnancy test(s) as verified by the Investigator. This applies even if the subject practices true abstinence from heterosexual contact.

    b. Either practice true abstinence from heterosexual contact or agree to use, and be able to comply with, effective measures of contraception without interruption.

    c. Agree to abstain from breastfeeding during study participation. d. Refrain from tissue donation including egg cell donation or any other tissue/blood/organ donations.
13. Male subjects must:

    a. Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, even if he has undergone a successful vasectomy.

    b. Refrain from tissue donation including sperm or any other tissue/blood/organ donations.
14. Only subjects that would be considered for any of the 5 proposed standard regimens (DPd, DVd, IRd, Kd, or EPd), as judged by the investigator, should be included in the study.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject has nonsecretory multiple myeloma (MM).
5. Subject has any of the following laboratory abnormalities:

   a. Absolute neutrophil count (ANC) < 1,000/μL b. Platelet count: < 75,000/μL in subjects in whom < 50% of bone marrow nucleated cells are plasma cells and platelet count < 50,000/μL in subjects in whom ≥ 50% of bone marrow nucleated cells are plasma cells (it is not permissible to transfuse a subject to reach this level) c. Hemoglobin < 8 g/dL (< 4.9 mmol/L) (it is not permissible to transfuse a subject to reach this level) d. Serum creatinine clearance (CrCl) < 45 mL/min e. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L) f. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN) g. Serum total bilirubin > 1.5 × ULN or > 3.0 mg/dL for subjects with documented Gilbert's syndrome h. International normalized ratio (INR) or activated partial thromboplastin time (aPTT) > 1.5 × ULN, or history of Grade ≥ 2 hemorrhage within 30 days, or subject requires ongoing treatment with chronic, therapeutic dosing of anticoagulants (eg, warfarin, low molecular weight heparin, Factor Xa inhibitors)
6. Subject has inadequate pulmonary function defined as oxygen saturation (SaO2) < 92% on room air.
7. Subject has prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years • Basal cell carcinoma of the skin

   • Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system) or prostate cancer that can be treated with curative intent
8. Subject has active or history of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome or amyloidosis.
9. Subject with known central nervous system (CNS) involvement with myeloma.
10. Subject has clinical evidence of pulmonary leukostasis and disseminated intravascular coagulation.
11. Subject has known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) 50% of predicted normal.
12. Subject has a history or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or other CNS bleed, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
13. Subject was treated with DARA in combination with POM with or without dex (DP±d) as part of their most recent anti-myeloma treatment regimen, cannot receive DPd as bridging therapy but may receive DVd, IRd, Kd or EPdas bridging as per Investigator's discretion if randomized to Treatment Arm A.
14. Subject was treated with DP±d as part of their most recent anti-myeloma treatment regimen, cannot receive DPd if randomized to Treatment Arm B but may receive DVd, IRd, Kd, or EPd as per Investigator's discretion.
15. Subject was treated with DARA in combination with BTZ with or without dexamethasone (DV±d) as part of their most recent anti-myeloma treatment regimen, cannot receive DVd as bridging therapy but may receive DPd, IRd, Kd, or EPd as bridging as per Investigator's discretion if randomized to Treatment Arm A.
16. Subject was treated with DV±d as part of their most recent anti-myeloma treatment regimen, cannot receive DVd if randomized to Treatment Arm B but may receive DPd, IRd, Kd, or EPd as per Investigator's discretion.
17. Subject was treated with IXA in combination with LEN with or without dexamethasone (IR±d) as part of their most recent anti-myeloma treatment regimen, cannot receive IRd as bridging therapy but may receive DPd, DVd, Kd, or EPd as bridging as per Investigator's discretion if randomized to Treatment Arm A.
18. Subject was treated with IR±d as part of their most recent anti-myeloma treatment regimen, cannot receive IRd if randomized to Treatment Arm B but may receive DPd, DVd, Kd, or EPd as per Investigator's discretion.
19. Previous history of an allogeneic hematopoietic stem cell transplantation, treatment with any gene therapy-based therapeutic for cancer, investigational cellular therapy for cancer or BCMA targeted therapy.
20. Subject has received autologous stem cell transplantation (ASCT) within 12 weeks prior to randomization.
21. Subject has received any of the following within the last 14 days prior to randomization:

    a. Plasmapheresis b. Major surgery (as defined by the Investigator) c. Radiation therapy other than local therapy for myeloma-associated bone lesions d. Use of any investigational agents and systemic anti-myeloma drug therapy
22. Echocardiogram (ECHO) or multigated acquisition (MUGA) with left ventricular ejection fraction (LVEF) < 45%.
23. Ongoing treatment with chronic immunosuppressants (eg, cyclosporine or systemic steroids at any dose). Intermittent topical, inhaled or intranasal corticosteroids are allowed.
24. Subject is positive for human immunodeficiency virus (HIV-1 and HIV-2), chronic or active hepatitis B or active hepatitis A or C.
25. Subject has uncontrolled systemic fungal, bacterial, viral or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antimicrobial treatment) or requiring IV antimicrobials for management.
26. Subject has a history of class III or IV congestive heart failure (CHF) or severe nonischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months prior to randomization.
27. Hypersensitivity to DARA, thalidomide, lenalidomide, POM, BTZ, IXA, CFZ, ELO or dexamathasone. This includes rash ≥ Grade 3 during prior thalidomide, POM or lenalidomide therapy.
28. Subject with known hypersensitivity to any component of bb2121 product, cyclophosphamide, fludarabine, and/or tocilizumab or hypersensitivity to the excipients contained in the formulation of DARA, POM, LEN, IXA, BTZ, CFZ, ELO or dexamethasone.
29. Subject is a female who is pregnant, nursing, or breastfeeding
30. For a subject randomized to Treatment Arm B and will be on a POM- or LEN-containing regimen; unable or unwilling to undergo protocol required thromboembolism prophylaxis.

28 Subject is intolerant to bortezomib, or has acute diffuse infiltrative pulmonary and pericardial disease, subject cannot receive DVd as bridging therapy if randomized to Treatment Arm A or cannot receive DVd if randomized to Treatment Arm B.

31. Subject was treated with K±d as part of their most recent anti-myeloma treatment regimen, cannot receive Kd if randomized to Treatment Arm B but may receive DPd, DVd, IRd or EPd as per Investigator's discretion.

32. Subject was treated with EP±d as part of their most recent anti-myeloma treatment regimen, cannot receive EPd if randomized to Treatment Arm B but may receive DPd, DVd, Kd or IRd as per Investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Minimum of 5 years from randomization
  Time from randomization to the first documentation of progressive disease based on the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma assessed by an independent response committee (IRC) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Minimum of 5 years from randomization
  Time from randomization to time of death due to any cause
Event-free Survival (EFS) | Minimum of 5 years from randomization
  Time from randomization to the first documentation of progressive disease, first day when subject receives another anti-myeloma treatment or death due to any cause, whichever occurs first
Overall Response Rate (ORR) | Minimum of 5 years from randomization
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by an IRC
Minimal Residual Disease (MRD) | Minimum of 5 years from randomization
  Percentage of MRD evaluable subjects that are MRD negative (defined at a minimum of 1 in 10^5 nucleated cells) using flow cytometry (EuroFlow) and next generation sequencing (NGS)
Complete Response (CR) Rate | Minimum of 5 years from randomization
  Percentage of subjects who achieved CR or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by an IRC
Duration of Response (DOR) | Minimum of 5 years from randomization
  Time from first documentation of response (PR or better) to first documentation of disease progression or death from any cause, whichever occurs first
Time to Response (TTR) | Minimum of 5 years from randomization
  TTR is calculated as the time from randomization to the initial documented response (PR or better) based on IMWG guideline for responders
Adverse Events (AEs) | Minimum of 5 years from randomization
  Number of participants with adverse events
Pharmacokinetics- Cmax | Minimum 5 years after bb2121 infusion
  Maximum peak in bb2121 chimeric antigen receptor (CAR) T cells
Pharmacokinetics- tmax | Minimum 5 years after bb2121 infusion
  Time to peak of bb2121 CAR T cells
Pharmacokinetics- AUC | Minimum 5 years after bb2121 infusion
  Area under the curve of CAR T cells
Pharmacokinetics- t-last | Minimum 5 years after bb2121 infusion
  Time to last measurable CAR T cells
Pharmacokinetics- AUC0-28days | Minimum 5 years after bb2121 infusion
  Area under the curve of CAR T cells from time zero to Day 28
Subject-reported outcomes as measured by European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC-QLQ-C30) | Minimum of 5 years from randomization
  Questionnaire will be used as a measure of health-related quality of life
Subject-reported outcomes as measured by EuroQoL Group European Quality of Life-5 Dimensions health state classifier to 5 Levels (EQ-5D-5L) Health Questionnaire | Minimum of 5 years from randomization
  Is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal
Subject-reported outcomes as measured by European Quality of Life Multiple Myeloma Module (EORTC-QLQ-MY20) | Minimum of 5 years from randomization
  Is a 20-item myeloma module intended for use among patients varying in disease stage and treatment modality
Time to next antimyeloma treatment | Minimum of 5 years from randomization
  Time from randomization to first day when subject receives another anti-myeloma treatment
Progression-free survival after next line therapy (PFS2) | Minimum of 5 years from randomization
  Time from randomization to second objective disease progression or death from any cause, whichever is first

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (34):
  - Local Institution - 109, Birmingham, Alabama
  - Local Institution - 141, Scottsdale, Arizona
  - Local Institution - 145, Los Angeles, California
  - Local Institution - 122, Los Angeles, California
  - Local Institution - 124, Palo Alto, California
  - Local Institution - 142, Aurora, Colorado
  - Local Institution - 108, Jacksonville, Florida
  - Local Institution - 102, Tampa, Florida
  - Local Institution - 131, Atlanta, Georgia
  - Local Institution - 140, Atlanta, Georgia
  - Local Institution - 139, Chicago, Illinois
  - Local Institution - 100, Indianapolis, Indiana
  - Local Institution - 112, Westwood, Kansas
  - Local Institution - 104, Baltimore, Maryland
  - Local Institution - 134, Boston, Massachusetts
  - Local Institution - 123, Boston, Massachusetts
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Local Institution - 125, Rochester, Minnesota
  - Local Institution - 114, St Louis, Missouri
  - Local Institution - 138, Hackensack, New Jersey
  - Local Institution - 119, New York, New York
  - Local Institution - 115, New York, New York
  - Local Institution - 135, New York, New York
  - Local Institution - 113, Durham, North Carolina
  - Local Institution - 111, Philadelphia, Pennsylvania
  - Local Institution - 110, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center William M. Cooper Ambulatory Care Pavillion, Pittsburgh, Pennsylvania
  - Local Institution - 106, Nashville, Tennessee
  - Local Institution - 118, Dallas, Texas
  - Local Institution - 103, Dallas, Texas
  - Local Institution - 132, Houston, Texas
  - Local Institution - 136, Salt Lake City, Utah
  - Local Institution - 105, Seattle, Washington
  - Local Institution - 107, Madison, Wisconsin
- Local Institution - 202, Leuven, Belgium
- Canada (2):
  - Local Institution - 302, Calgary, Alberta
  - Local Institution - 303, Toronto, Ontario
- France (4):
  - Local Institution - 402, Lille
  - Local Institution - 403, Nantes
  - Local Institution - 400, Paris
  - Local Institution - 401, Toulouse
- Germany (5):
  - Local Institution - 515, Cologne
  - Local Institution - 513, Düsseldorf
  - Local Institution - 514, Hamburg
  - Local Institution - 512, Heidelberg
  - Local Institution - 511, Würzburg
- Local Institution - 611, Bologna, Italy
- Japan (4):
  - Local Institution - 806, Bunkyō City
  - Local Institution - 804, Isehara City, Kanagawa
  - Local Institution - 807, Nagoya
  - Local Institution - 805, Shibuya-ku
- Netherlands (2):
  - Local Institution - 650, Amsterdam
  - Local Institution - 651, Rotterdam
- Local Institution - 700, Oslo, Norway
- Spain (2):
  - Local Institution - 750, Pamplona
  - Local Institution - 751, Salamanca
- Local Institution - 800, Stockholm, Sweden
- Local Institution - 251, Bern, Switzerland
- United Kingdom (2):
  - Local Institution - 850, Leeds
  - Local Institution - 851, London

REFERENCES:
- [Derived] Lopez-Munoz N, Bar N, Diels J, van Sanden S, Mendes J, Lee S, Hernando T, Lendvai N, Patel N, Ishida T, Er J, Harrison SJ. Ciltacabtagene Autoleucel Versus Idecabtagene Vicleucel in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma with 2-4 Prior Lines of Therapy: Updated Matching-Adjusted Indirect Comparison. Adv Ther. 2026 Feb 2. doi: 10.1007/s12325-025-03479-y. Online ahead of print. PMID 41627370
- [Derived] Ailawadhi S, Arnulf B, Patel K, Cavo M, Nooka AK, Manier S, Callander N, Costa LJ, Vij R, Bahlis NJ, Moreau P, Solomon S, Abrahamsen IW, Baz R, Broijl A, Chen C, Jagannath S, Raje N, Scheid C, Delforge M, Benjamin R, Pabst T, Iida S, Berdeja J, Giralt S, Truppel-Hartmann A, Chen Y, Zhong X, Wu F, Piasecki J, Eliason L, Dhanda D, Felten J, Caia A, Cook M, Popa McKiver M, Rodriguez-Otero P. Ide-cel vs standard regimens in triple-class-exposed relapsed and refractory multiple myeloma: updated KarMMa-3 analyses. Blood. 2024 Dec 5;144(23):2389-2401. doi: 10.1182/blood.2024024582. PMID 39197072
- [Derived] Rodriguez-Otero P, Ailawadhi S, Arnulf B, Patel K, Cavo M, Nooka AK, Manier S, Callander N, Costa LJ, Vij R, Bahlis NJ, Moreau P, Solomon SR, Delforge M, Berdeja J, Truppel-Hartmann A, Yang Z, Favre-Kontula L, Wu F, Piasecki J, Cook M, Giralt S. Plain language summary of the KarMMa-3 study of ide-cel or standard of care regimens in people with relapsed or refractory multiple myeloma. Future Oncol. 2024;20(18):1221-1235. doi: 10.2217/fon-2023-0954. Epub 2024 Apr 23. PMID 38651976
- [Derived] Rodriguez-Otero P, Ailawadhi S, Arnulf B, Patel K, Cavo M, Nooka AK, Manier S, Callander N, Costa LJ, Vij R, Bahlis NJ, Moreau P, Solomon SR, Delforge M, Berdeja J, Truppel-Hartmann A, Yang Z, Favre-Kontula L, Wu F, Piasecki J, Cook M, Giralt S. Ide-cel or Standard Regimens in Relapsed and Refractory Multiple Myeloma. N Engl J Med. 2023 Mar 16;388(11):1002-1014. doi: 10.1056/NEJMoa2213614. Epub 2023 Feb 10. PMID 36762851
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome